CLINICAL TRIAL: NCT00467909
Title: Efficacy of Fortified Products on Improving Long Term Cognitive Performance in School Children in India
Brief Title: Nutrition and Cognition in Indian Children
Acronym: CHAMPION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. John's Research Institute (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 04B9-P
Record Dates: First submitted 2007-04-30; First posted 2007-05-01 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2007-04

CONDITIONS: Healthy
Keywords: micronutrients; cognition; DHA; healthy children
MeSH Terms: interventions — Micronutrients

STUDY DESIGN:
Intervention Model Description: In a 2-by-2 factorial, double-blind, randomized controlled trial, 598 children aged 6-10 y were individually allocated to 1 of 4 intervention groups to receive foods fortified with either 100% or 15% of the Recommended Dietary Allowance of micronutrients in combination with either 900 mg α-linolenic acid plus 100 mg docosahexaenoic acid or 140 mg α-linolenic acid for 12 mo. Anthropometric and biochemical assessments were performed at baseline and 12 mo. Cognitive performance was measured at baseline and at 6 and 12 mo.
Who Masked: Participant, Care Provider
Masking Description: The drink (nutritional item) was prepared daily, for each child individually, by mixing 65 g of the powder in 160 mL boiled water. The fortified products in the 4 treatment groups were each assigned a specific color code, which was displayed on the package, but were otherwise indistinguishable in color, appearance, and taste. The investigators, assessors of cognitive tests, and participants were blinded until the study was completed, all data were entered, and the initial analyses were performed.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Hgh micronutrients, high n-3 fatty acid treatment Arm (Experimental): High micronutrients, high n-3 fatty acid treatment The high micronutrient treatment provided 100% of the RDA of iodine, iron, riboflavin, vitamin B-6, vitamin B-12, folate, and vitamin A for children 7-9 y of age (25) (Table 1). To optimize the bioavailability of iron, zinc was provided at 92% of the RDA based on a molar ratio of 2 (iron) to 1 (zinc), vitamin C was provided at 650% of the RDA based on a molar ratio of 4 (vitamin C) to 1 (iron) and, calcium was provided at 33% of the RDA to minimize possible inhibition of iron absorption (26., 27., 28.).
  Interventions: Behavioral: micronutrients
- low micronutrients, high n-3 fatty acid treatment (Experimental): low micronutrients, high n-3 fatty acid treatment The low micronutrient treatment delivered micronutrients per kcal proportional to that consumed by the children in their habitual diet (S Muthayya, 2006, unpublished observations). This amounted to 15% of the RDA provided in 420 kcal. The high n-3 treatment provided 900 mg ALA, which is 50% of the recommended intake of ALA for children aged 2-12 y (29), and 100 mg DHA, which corresponds with ≈50% of the recommended fish intake for children
  Interventions: Behavioral: micronutrients
- low micronutrients, low n-3 fatty acid treatment. (Experimental): low micronutrients, low n-3 fatty acid treatment. The low micronutrient treatment delivered micronutrients per kcal proportional to that consumed by the children in their habitual diet (S Muthayya, 2006, unpublished observations). This amounted to 15% of the RDA provided in 420 kcal. The high n-3 treatment provided 900 mg ALA, which is 50% of the recommended intake of ALA for children aged 2-12 y (29), and 100 mg DHA, which corresponds with ≈50% of the recommended fish intake for children
  Interventions: Behavioral: micronutrients
- high micronutrients, low n-3 fatty acid treatment (Experimental): high micronutrients, low n-3 fatty acid treatment The high micronutrient treatment provided 100% of the RDA of iodine, iron, riboflavin, vitamin B-6, vitamin B-12, folate, and vitamin A for children 7-9 y of age (25) (Table 1). To optimize the bioavailability of iron, zinc was provided at 92% of the RDA based on a molar ratio of 2 (iron) to 1 (zinc), vitamin C was provided at 650% of the RDA based on a molar ratio of 4 (vitamin C) to 1 (iron) and, calcium was provided at 33% of the RDA to minimize possible inhibition of iron absorption (26., 27., 28.).
  Interventions: Behavioral: micronutrients

INTERVENTIONS:
Behavioral: micronutrients

SUMMARY:
Nutritional deficiencies are a major problem in school children in India and have a variety of adverse effects on their cognitive development and growth, and increase susceptibility to infections. There is strong evidence for beneficial effects of iodine, iron and protein-energy on cognitive development in children, while evidence for vitamin B6, vitamin B12, folate, zinc and, omega-3 fatty acids and in particular docosahexanoic acid (DHA) is limited and inconclusive. A randomised, double-blind, placebo-controlled 2x2 factorial design will be conducted to assess the effect of a micronutrient with or without omega-3 fatty acids on cognitive development and performance and other selected outcome variables such as growth, morbidity and immune response in children of 7-9 years of age in India.

DETAILED DESCRIPTION:
Nutritional deficiencies are a major problem in school children in India and have a variety of adverse effects on their cognitive development and growth, and increase susceptibility to infections. There is strong evidence for beneficial effects of iodine, iron and protein-energy on cognitive development in children, while evidence for vitamin B6, vitamin B12, folate, zinc and, omega-3 fatty acids and in particular docosahexanoic acid (DHA) is limited and inconclusive. The present study will investigate the efficacy of foods fortified with omega-3 fatty acids including DHA and a micronutrient mix (iodine, iron, vitamin B2, vitamin B6, vitamin B12, folate, zinc, calcium, vitamin A, vitamin C and vitamin E) on improving cognitive development and performance in school children in India.

The study will follow a randomised, double-blind, placebo-controlled 2x2 factorial design in which children aged 7-9 years will be randomised to one of four treatment groups and prospectively followed for a period of twelve months to assess cognitive development and performance and other selected outcome variables such as growth, morbidity and immune response. Intervention will take place in primary schools, where children will receive three intervention products daily. The products will contain omega-3 fatty acids with micronutrients, or micronutrients only, or omega3 fatty acids only or a placebo. At baseline, 6 and 12 months cognitive tests will be administered and blood samples will be drawn to assess nutritional status and immune response to hepatitis B vaccination. Compliance will be measured daily and morbidity will be monitored weekly by means of a questionnaire. Anthropometric measurements will be carried out monthly.

It is expected that, after 12 months of intervention, children consuming products containing omega-3 fatty acids with micronutrients will have statistically significant higher scores and higher improvement in scores on cognitive tests, will grow taller and have a better immune response than children consuming control products.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 7to 9 years, not having their tenth birthday close to the start of the study
2. Children attending the primary schools in Bangalore area in India which are selected in the cross-sectional survey
3. Healthy as assessed by a physician
4. Willing to consume the test product
5. Willing to participate in the study and perform all measurements including cognitive testing, blood drawing, urine samples, anthropometry, dietary intake and questionnaires.
6. Informed consent signed by parent or caregiver and oral consent given by child
7. Parents intend to stay in the study area for less than 1 year.

Exclusion Criteria:

1. Children with obvious mental and physical handicaps
2. Children using medication which interferes with study measurements
3. Reported dietary restrictions such as a medically prescribed diet, or a slimming diet prior to or during the study
4. Severely undernourished as defined by HAZ, WAZ or WHZ greater than -3 SD from NCHS reference standard z-scores (Ogden et al, 2002)
5. Severely iron deficient as defined by hemoglobin concentrations <80 g/L (WHO, 2001)
6. Reported participation in another biomedical trial 3 months before the start of the study or during the study.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2005-11-01 (Actual); Primary Completion 2007-03-31 (Actual); Study Completion 2007-03-31 (Actual)

PRIMARY OUTCOMES:
Cognitive development and performance | 1 year
  Cognitive performance was measured at baseline and at 6 and 12 mo.

SECONDARY OUTCOMES:
Growth, Morbidity, Immune function and gut function | 1 year
  Weight, height (linear growth), and MUAC after 12 mo of interventionwith baseline values

CONTACTS AND LOCATIONS:
Overall Officials: Anura V Kurpad, MD, Principal Investigator — St. John's Research Institute
Locations (1):
- St John's research Institute, Bangalore, Karnataka, India

REFERENCES:
- [Result] Muthayya S, Eilander A, Transler C, Thomas T, van der Knaap HC, Srinivasan K, van Klinken BJ, Osendarp SJ, Kurpad AV. Effect of fortification with multiple micronutrients and n-3 fatty acids on growth and cognitive performance in Indian schoolchildren: the CHAMPION (Children's Health and Mental Performance Influenced by Optimal Nutrition) Study. Am J Clin Nutr. 2009 Jun;89(6):1766-75. doi: 10.3945/ajcn.2008.26993. Epub 2009 Apr 15. PMID 19369376